CLINICAL TRIAL: NCT00367419
Title: Low-Dose Long-Term Prescription of Erythromycin in Mustard-Induced Bronchiolitis Obliterans
Brief Title: Use of Erythromycin in Mustard-Induced Bronchiolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: S-340-14-6-1-PU-02
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2006-03

CONDITIONS: Bronchiolitis Obliterans; Acute Obliterating Bronchiolitis
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Erythromycin

INTERVENTIONS:
Drug: Erythromycin

SUMMARY:
We looked for the effectiveness of low-dose long-term prescription of erythromycin in mustard-induced bronchiolitis obliterans

ELIGIBILITY:
Inclusion Criteria:

* Documented chemical exposure
* Clinical, spirometric and radiological findings were compatible with BO on High Resolution Computed Tomography (HRCT)
* Non-responsiveness to high dose bronchodilator therapy

Exclusion Criteria:

* Radiographic evidence of pneumonia, active tuberculosis, lung carcinoma, or an infection that necessitated the use of an antibiotic
* History of cigarette smoking and occupational exposure to toxic agents of hypersensitivity to macrolides
* History of treatment with a systemic antibiotic within 7 days before the start of the study
* Any investigational medicine within 4 weeks of the study
* History of antibiotic injection within 6 weeks before the study
* Concomitant Theophylline or Carbamazepine, unless their serum concentrations were regularly monitored
* Patients who were in the exacerbation phase of their respiratory complications
* Need to use medications interact with macrolides such as Digoxin, Theophylline and Carbamazepine
* Systemic antibiotics
* Systemic Corticosteroids
* Admission to the hospital
* Abnormal kidney or liver function

Sex: Male
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ghanei, Professor, Study Director — Research Center of Chemical Injuries, Baqyatallah Medical Sciences University, Tehran, Iran
Locations (1):
- Baqiyatallah Medical Sciences University, Tehran, Tehran Province, Iran